CLINICAL TRIAL: NCT02430168
Title: Comparison of RIRS Versus PCNL Methods, According to Postoperative Pain and Analgesic Demand in 2 to 4 cm Renal Stones
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, Nihat Karakoyunlu, MD, Diskapi Teaching and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2-4 cm RIRS vs PCNL
Record Dates: First submitted 2015-04-22; First posted 2015-04-30 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2015-04

CONDITIONS: Kidney Stones
Keywords: Stone; RIRs; PCNL; Pain
MeSH Terms: conditions — Kidney Calculi; Calculi; Pain | interventions — Nephrolithotomy, Percutaneous

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- RIRS (Active Comparator): Retrograde intrarenal surgery
  Interventions: Procedure: Retrograde intrarenal surgery
- PCNL (Active Comparator): Percutaneous nephrolithotomy
  Interventions: Procedure: Percutaneous nephrolithotomy

INTERVENTIONS:
Procedure: Percutaneous nephrolithotomy
  Other Names: PCNL
  Arms: PCNL
Procedure: Retrograde intrarenal surgery
  Other Names: RIRS
  Arms: RIRS

SUMMARY:
Purpose: to investigate the postoperative outcomes of Retrograde intrarenal surgery versus percutaneous nephrolithotomy in 2 to 4 cm kidney stones.

ELIGIBILITY:
Inclusion Criteria:

* The patients who have 2 to 4 cm kidney stones
* ASA score within 1 to 3

Exclusion Criteria:

* Previous surgical treatment including SWL
* Congenital abnormalities

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-12; Primary Completion 2016-12 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Analgesic demand | Postoperative 24 hours
Stone clearance | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Diskapi TRH, Ankara, Turkey (Türkiye)

REFERENCES:
- [Result] Akman T, Binbay M, Ozgor F, Ugurlu M, Tekinarslan E, Kezer C, Aslan R, Muslumanoglu AY. Comparison of percutaneous nephrolithotomy and retrograde flexible nephrolithotripsy for the management of 2-4 cm stones: a matched-pair analysis. BJU Int. 2012 May;109(9):1384-9. doi: 10.1111/j.1464-410X.2011.10691.x. Epub 2011 Oct 28. PMID 22093679
- [Derived] Soderberg L, Ergun O, Ding M, Parker R, Borofsky MS, Pais V, Dahm P. Percutaneous nephrolithotomy versus retrograde intrarenal surgery for treatment of renal stones in adults. Cochrane Database Syst Rev. 2023 Nov 13;11(11):CD013445. doi: 10.1002/14651858.CD013445.pub2. PMID 37955353